CLINICAL TRIAL: NCT03761862
Title: Evaluation of the Neural Therapy Effect on Long Term Postoperative Discomforts and Gynecologic Symptoms in Patients
Brief Title: Evaluation of the Neural Therapy Effect on Long Term Postoperative Discomforts in Patients Who Undergo Bilateral Tubal Ligation
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: Neuraltherapyinbtl
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Pain, Postoperative; Neural Therapy of Huneke; Dysmenorrhea; Dyspareunia; Sterilization, Tubal
MeSH Terms: conditions — Pain, Postoperative; Dysmenorrhea; Dyspareunia | interventions — Anesthesia, Local

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: The control group with bilateral tubal ligation
  Interventions: Procedure: Neural Therapy
- Neural Therapy: The treatment group
  Interventions: Procedure: Neural Therapy

INTERVENTIONS:
Procedure: Neural Therapy — Neural therapy is a form of alternative medicine in which local anesthetic is injected into certain locations of the body in an attempt to treat chronic pain and illness.

SUMMARY:
The aim of this study was to explore the effect of neural therapy on postoperative pain and discomfort such as abdominal swelling; and gynecologic symptoms such as dysmenorrhea, dyspareunia, amount of menstrual bleeding and vaginitis. It also aimed to find out any possible links between the clinical changes and pathophysiologic mechanisms. One hundred and thirteen patients were randomly divided into two groups (neural therapy and control). Postoperative first day, neural therapy was applied to the T10 to S4 dermatomes and utero-vaginal ganglion in random with local anesthetic agent. All patients were recalled one year after the treatment. The visual analog scale (VAS) were noted in both groups, also discomfort and gynecologic symptoms are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo bilateral tubal ligation

Exclusion Criteria:

* Previous abdominal surgery
* Patients with diseases that could have neurologic complications (DM, SLE ...)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who undergo bilateral tubal ligation admitted to the training and research hospital.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Pain scores | 1 year later
  Visual Analog Scale was used as the pain scale.1 to 10 points are given here. High score (8- 10) indicates severe pain.